CLINICAL TRIAL: NCT06619067
Title: Efficacy Study of the Probiotic Food Supplement PROBAFLOR for Maintaining Intestinal Well-being: Single-centre, Controlled, Randomized, Parallel Group, Double-blind Clinical Study
Brief Title: Efficacy Study of the Probiotic Food Supplement PROBAFLOR for Maintaining Intestinal Well-being
Acronym: PROBAFLOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synbiotec Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024/19
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Gut; Microbiota Balance
Keywords: Probiotics; Gut health; Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated group (Active Comparator): Dietary supplement: PROBAFLOR 20 Billion CFU/dose, serving size = 1 capsule/day
  Interventions: Dietary Supplement: PROBAFLOR
- Placebo group (Placebo Comparator): Placebo Placebo product, serving size = 1 capsule/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: PROBAFLOR — PROBAFLOR is a food supplement made up of 11 bacterial strains and inulin. The bacterial strains present are: Bifidobacterium lactis BLC1, Lactococcus lactis LL82, Lactobacillus plantarum 14D, Lactobacillus acidophilus LA1, Streptococcus thermophilus Z57, Bifidobacterium longum SP54, Lactobacillus rhamnosus SP1, Lactobacillus bulgaricus LB2, Bifidobacterium bifidum SP9,Lactobacillus salivarius SP2, Lactobacillus casei BGP93.
  Arms: Treated group
Other: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
It is now known that intestinal health has a strong influence on the entire body. Recent research advances have demonstrated the involvement of the intestinal microbiota in the well-being of the intestine. Preventive medicine is increasingly perceived as important in medical and economic terms, particularly in the field of gastroenterology. An innovative approach to support gut health is based on the use of modulators of the intestinal microbiome or gastrointestinal barrier, such as probiotics or prebiotics. The rationale for this study is therefore based on the hypothesis that the combination of 11 probiotic strains, conveyed through the PROBAFLOR food supplement, can play a positive role in maintaining normal intestinal function, bringing benefits to the subject who takes this supplement.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled intervention study with a duration of 3 months of intervention + 1 month of follow-up, on biological samples. Eligible participants will be randomized and receive either the probioic or placebo supplement to consume daily for 3 months. Three check-in visits will occur, one at the screening, the second one afetr the 3-months intervention and the final one after 1 month of followup. Participants will be expected to complete a daily study diary documenting their investigational product use/adverse events and a daily bowel habits diary documenting each bowel movement. Stool samples, and questionnaires will be completed for study outcome analysis.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 18 and 65;
* healthy based on medical history;
* commitment to comply with all firm procedures;
* commitment to refrain from using any home remedies to control gastrointestinal problems, particularly if live bacteria are involved;
* signature of informed consent.

Exclusion Criteria:

* use of probiotics continuously, in the two months prior to enrollment;
* use of antibiotics in the month before enrollment;
* chemotherapy treatments;
* diagnosis of respiratory, hepatic and/or renal failure;
* Clinically significant diseases of the gastrointestinal tract (examples include, but are not limited to, celiac disease, gluten intolerance/sensitivity, inflammatory bowel disease);
* Women who are pregnant, breastfeeding or planning to become pregnant during the study;
* Allergy or sensitivity to the active or inactive ingredients of the investigational product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
maintenance and/or improvement of intestinal health and health-related quality of life (through the GIQLI questionnaire) | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration

SECONDARY OUTCOMES:
Intestinal microbiota composition | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration
  Metagenomic analysis on faecal samples
SCFA determination | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration
  Gas chromatographic analysis of fecal water
Changes in quality of life. | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration
  Assessed by PGWBI (The Psychological General Well-Being Index)
Changes in intestinal functionality | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration
  Assessed in accordance with the Bristol Stool Form Scale
Changes on gastrointestinal symptoms | Baseline, After 3 months of intervention, at follow-up (one month after the end of administration
  Assessed by the GSRS (Gastrointestinal Symptom Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Verdenelli, PhD, Study Director — Synbiotec Srl
Locations (1):
- Scuola di Bioscienze e Medicina Veterinaria, Università di Camerino, Camerino, Macerata, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Revicki DA, Wood M, Wiklund I, Crawley J. Reliability and validity of the Gastrointestinal Symptom Rating Scale in patients with gastroesophageal reflux disease. Qual Life Res. 1998 Jan;7(1):75-83. doi: 10.1023/a:1008841022998. PMID 9481153
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Sanchez B, Delgado S, Blanco-Miguez A, Lourenco A, Gueimonde M, Margolles A. Probiotics, gut microbiota, and their influence on host health and disease. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600240. Epub 2016 Oct 10. PMID 27500859
- [Background] Possemiers S, Grootaert C, Vermeiren J, Gross G, Marzorati M, Verstraete W, Van de Wiele T. The intestinal environment in health and disease - recent insights on the potential of intestinal bacteria to influence human health. Curr Pharm Des. 2009;15(18):2051-65. doi: 10.2174/138161209788489159. PMID 19519443
- [Background] Mai V, Morris JG Jr. Colonic bacterial flora: changing understandings in the molecular age. J Nutr. 2004 Feb;134(2):459-64. doi: 10.1093/jn/134.2.459. PMID 14747689
- [Background] Tuohy KM, Probert HM, Smejkal CW, Gibson GR. Using probiotics and prebiotics to improve gut health. Drug Discov Today. 2003 Aug 1;8(15):692-700. doi: 10.1016/s1359-6446(03)02746-6. PMID 12927512
- [Background] Sola KF, Vladimir-Knezevic S, Hrabac P, Mucalo I, Saso L, Verbanac D. The effect of multistrain probiotics on functional constipation in the elderly: a randomized controlled trial. Eur J Clin Nutr. 2022 Dec;76(12):1675-1681. doi: 10.1038/s41430-022-01189-0. Epub 2022 Aug 4. PMID 35927504
- [Background] Rizzardini G, Eskesen D, Calder PC, Capetti A, Jespersen L, Clerici M. Evaluation of the immune benefits of two probiotic strains Bifidobacterium animalis ssp. lactis, BB-12(R) and Lactobacillus paracasei ssp. paracasei, L. casei 431(R) in an influenza vaccination model: a randomised, double-blind, placebo-controlled study. Br J Nutr. 2012 Mar;107(6):876-84. doi: 10.1017/S000711451100420X. Epub 2011 Sep 7. PMID 21899798